CLINICAL TRIAL: NCT02100020
Title: A Community-based Randomized Controlled Trial Testing Implementation of the New Canadian Physical Activity Guidelines for Adults With Multiple Sclerosis.
Brief Title: Implementing Physical Activity Guidelines for Adults With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MSProject2001
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: physical activity; exercise guidelines; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Referral to Physical Activity (Experimental): The REF group will be referred to a centre-based community exercise program in their respective community (either the MacWheelers or Revved Up) by a clinical neurologist where they will be prescribed exercise based on the PAGs for adults with MS, and according to their individual capabilities.
  Interventions: Other: Direct Referral to physical activity
- Control (No Intervention): The CON group will be provided with a print copy of the PAGs and a link to an online resource for physical activity information.

INTERVENTIONS:
Other: Direct Referral to physical activity — Participants randomized to the Direct Referral to Physical Activity Arm will be provided with a referral to a physical activity program in their community and will be closely monitored in this program for 16 wks.
  Arms: Direct Referral to Physical Activity

SUMMARY:
The proposed project will evaluate two methods of implementation of the new Physical Activity Guidelines (PAGs) for Adults with Multiple Sclerosis (MS) living in two Ontario communities. The investigators will also determine if following the PAGs will improve aspects of fitness, function, quality of life and risk for cardiometabolic disease in this population. The investigators hypothesize that adherence to the PAGs will be higher in people who have been referred directly to a community-based exercise program, and that this greater adherence to physical activity will be associated with greater improvements in fitness, function and quality of life.

This randomized controlled trial will provide important information on how best to implement physical activity recommendations within the community setting; this information will be translated to key stakeholders during the final stages of the project.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS with mild-moderate disability (EDSS 1-7)
* Aged 18-60
* Medical clearance to participate in physical activity

Exclusion Criteria:

* current participation in regular physical activity (at least twice-weekly)
* other serious medical condition that might impair ability to participate in strength or aerobic exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the Physical Activity Guidelines | 3 years
  Adherence to the physical activity guidelines will be analyzed by having participants fill in a weekly physical activity log that will be sent to them by email.

SECONDARY OUTCOMES:
Physical Fitness | At baseline and after the 16 week intervention
  Peak oxygen uptake, maximum muscle strength, bodyweight
Perceived Quality of Life | At baseline and after the 16 week intervention
  Multiple Sclerosis Quality of Life (MSQoL) scale
Fatigue | At baseline and after the 16 week intervention
  Multiple Sclerosis Fatigue Impact Scale (MSFIS)
Mobility | At baseline and after the 16 week intervention
  25ft walk test
Blood markers of cardiovascular disease risk | At baseline and after the 16 week intervention
  blood lipid panel, HbA1c, fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L Hicks, Ph.D., Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster University, Physical Activity Centre for Excellence, Hamilton, Ontario
  - Queens University, Kingston, Ontario

REFERENCES:
- [Derived] Canning KL, Hicks AL. Physician referral improves adherence to the physical activity guidelines for adults with MS: A randomized controlled trial. Mult Scler Relat Disord. 2020 Jan;37:101441. doi: 10.1016/j.msard.2019.101441. Epub 2019 Oct 22. PMID 31675636